CLINICAL TRIAL: NCT04814433
Title: A Randomized, Single-Blinded, Placebo-Controlled Study Evaluating Postoperative Non-Opioid Pain Management Utilizing Local Anesthetics Coupled With Modulated Coagulation
Brief Title: Evaluating Postoperative Non-Opioid Pain Management Utilizing Local Anesthetics Coupled With Modulated Coagulation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Both lack of enrollment as well as study staff turnover
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-01420
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Opioid Pain Medication
MeSH Terms: interventions — Tranexamic Acid; Aminocaproic Acid; recombinant human thrombin; Lidocaine; Epinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Topical lidocaine and bupivacaine alone (Experimental): In this treatment group, each solution will include 5 ml of 1% lidocaine, 5 ml of 0.25% bupivacaine
  Interventions: Drug: Lidocaine Hydrochloride with Epinephrine; Drug: Bupivacaine Hydrochloride with Epinephrine
- Topical lidocaine and bupivacaine with thrombin (Experimental): In this treatment group, each solution will include 5 ml of 1% lidocaine, 5 ml of 0.25% bupivacaine, 10000 units of thrombin
  Interventions: Drug: Recombinant Human Thrombin; Drug: Lidocaine Hydrochloride with Epinephrine; Drug: Bupivacaine Hydrochloride with Epinephrine
- Topical lidocaine and bupivacaine with thrombin and tranexamic acid (Experimental): In this treatment group, each solution will include 5 ml of 1% lidocaine, 5 ml of 0.25% bupivacaine, 10000 units of thrombin, and 500 mg of tranexamic acid
  Interventions: Drug: Tranexamic acid; Drug: Recombinant Human Thrombin; Drug: Lidocaine Hydrochloride with Epinephrine; Drug: Bupivacaine Hydrochloride with Epinephrine
- Topical lidocaine and bupivacaine with thrombin and aminocaproic acid (Experimental): In this treatment group, each solution will include 5 ml of 1% lidocaine, 5 ml of 0.25% bupivacaine, 10000 units of thrombin, and 1000 mg of aminocaproic acid
  Interventions: Drug: Tranexamic acid; Drug: Aminocaproic acid; Drug: Recombinant Human Thrombin; Drug: Lidocaine Hydrochloride with Epinephrine; Drug: Bupivacaine Hydrochloride with Epinephrine

INTERVENTIONS:
Drug: Tranexamic acid — FDA-approved usage for intravenous tranexamic acid (TXA) is for heavy menstrual bleeding and short-term prevention in patients with hemophilia.
  Total dose of 500 mg (20 mL) total will be given.
  Arms: Topical lidocaine and bupivacaine with thrombin and aminocaproic acid; Topical lidocaine and bupivacaine with thrombin and tranexamic acid
Drug: Aminocaproic acid — FDA notes that aminocaproic acid is useful in enhancing hemostasis when fibrinolysis contributes to bleeding. Aminocaproic acid inhibits both the action of plasminogen activators and to a lesser degree, plasmin activity. The fibrinolysis-inhibitory effects of aminocaproic acid appear to be exerted principally via inhibition of plasminogen activators and to a lesser degree through antiplasmin activity. Parenteral drug products should be inspected visually for particulate matter and discoloration prior to administration, whenever solution and container permit.
  Total of 1000 mg total will be given.
  Arms: Topical lidocaine and bupivacaine with thrombin and aminocaproic acid
Drug: Recombinant Human Thrombin — Topical thrombin is FDA approved as an aid to hemostasis whenever oozing blood and minor bleeding from capillaries and small venules is accessible and control of bleeding by standard surgical techniques is not sufficient.
  Recombinant human thrombin is available as 5000-unit and 20,000-unit vials of sterile recombinant topical thrombin lyophilized powder for solution. When reconstituted as directed, the final solution contains 1000 units/mL.
  For topical application, a total of 10000 units per open surgical study arm involving use of Thrombin will be given
  Arms: Topical lidocaine and bupivacaine with thrombin; Topical lidocaine and bupivacaine with thrombin and aminocaproic acid; Topical lidocaine and bupivacaine with thrombin and tranexamic acid
Drug: Lidocaine Hydrochloride with Epinephrine — Topical lidocaine product is FDA approved as an amide local anesthetic in any indication for relief of pain associated with superficial minor surgery and as an adjunct for local infiltration anesthesia. It is frequently used as a standard local anesthetic for surgical procedures.
  Each mL contains lidocaine hydrochloride and epinephrine, with 0.5 mg sodium metabisulfite as an antioxidant and 0.2 mg citric acid as a stabilizer.
  Total of 5 mLs per open surgical study arm involving lidocaine hydrochloride and epinephrine will be given
Drug: Bupivacaine Hydrochloride with Epinephrine — Topical bupivacaine is FDA approved as indicated for the production of local anesthesia for procedures by infiltration injection. It is frequently used as a standard local anesthetic for surgical procedures.
  Each mL contains bupivacaine hydrochloride and 0.005 mg epinephrine, with 0.5 mg sodium metabisulfite as an antioxidant and 0.2 mg citric acid (anhydrous) as stabilizer.
  Total of 5 mLs per open surgical study arm involving Bupivacaine Hydrochloride with Epinephrine will be given

SUMMARY:
This study is a prospective randomized trial examining the effect of topically combined antifibrinolytics (Tranexamic acid) with local anesthetics in all electively created surgical wound beds in hand surgery to provide long term pain relief and decrease the use of postoperative narcotics.

DETAILED DESCRIPTION:
The aim of the study is to provide long term pain relief and decrease the use of postoperative narcotics. All treatments are applied topically to the surgical bed prior to closure of the skin. Each of the drugs used in this study are Food and Drug Administration (FDA) approved and routinely used for pain relief. However, the route of administration of the drugs and addition of tranexamic acid or aminocaproic acid is considered off-label (outside of the FDA-approved indications) and therefore investigational.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Any patient undergoing elective hand surgery

Exclusion Criteria:

* Any patient with a traumatic open wound (only surgically created wounds will be included)
* History of chronic pain
* History of narcotic addiction
* History of recreational drug dependency
* History of psychiatric pathology
* Allergy to local anesthetics, recombinant human thrombin or tranexamic acid
* Any patient receiving a supra/infraclavicular block for anesthesia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chiu, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Thomas.Calahan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical Lidocaine and Bupivacaine Alone | Topical Lidocaine and Bupivacaine With Thrombin | Topical Lidocaine and Bupivacaine With Thrombin and Tranexamic Acid | Topical Lidocaine and Bupivacaine With Thrombin and Aminocaproic Acid
Started | 12 | 14 | 9 | 11
Completed | 8 | 6 | 5 | 6
Not Completed | 4 | 8 | 4 | 5
Not completed — Survey not returned | 4 | 8 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Lidocaine and Bupivacaine Alone | Topical Lidocaine and Bupivacaine With Thrombin | Topical Lidocaine and Bupivacaine With Thrombin and Tranexamic Acid | Topical Lidocaine and Bupivacaine With Thrombin and Aminocaproic Acid | Total
Number analyzed (Participants) | 8 | 6 | 5 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (2.7) | 57 (3.2) | 61 (2.8) | 53 (3.4) | 56 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 5 | 19
  Male | 2 | 2 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 0 | 2 | 9
  Not Hispanic or Latino | 2 | 3 | 5 | 4 | 14
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 1 | 4
  White | 2 | 2 | 3 | 3 | 10
  More than one race | 4 | 3 | 0 | 2 | 9
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 5 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Postoperative Pain Control
Description: Measured by self-reported level of pain recorded in a daily pain diary made by the researchers from the day of the surgery until post-operative day 14. The levels of pain are scored in the following manner: 1-2 no pain, 3-4 mild pain, 5-6 moderate pain, 7-8 severe pain, 9-10 worst pain imaginable.
Time Frame: Day 1 preoperative , Day 14 postoperative
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Topical Lidocaine and Bupivacaine Alone | Topical Lidocaine and Bupivacaine With Thrombin | Topical Lidocaine and Bupivacaine With Thrombin and Tranexamic Acid | Topical Lidocaine and Bupivacaine With Thrombin and Aminocaproic Acid
Number analyzed (Participants) | 8 | 6 | 5 | 6
units on a scale | 4.8 [3 to 8] | 4.4 [4 to 5] | 5.1 [2 to 7] | 4.7 [3 to 7]

2. Secondary Outcome: Amount of Opioid Pain Medication Required Postoperatively
Description: Measured by self-reported number of pain pills taken postoperatively until post-operative day 14.
Time Frame: From Day 1 postoperative to Day 14 postoperative
Measure: Mean (Full Range); unit: Pills
Arm/Group | Topical Lidocaine and Bupivacaine Alone | Topical Lidocaine and Bupivacaine With Thrombin | Topical Lidocaine and Bupivacaine With Thrombin and Tranexamic Acid | Topical Lidocaine and Bupivacaine With Thrombin and Aminocaproic Acid
Number analyzed (Participants) | 8 | 6 | 5 | 6
Pills | 5.5 [1 to 9] | 5 [2 to 8] | 5.7 [1 to 10] | 6 [2 to 9]

3. Secondary Outcome: Total Time in Post Anesthesia Care Unit (PACU)
Time Frame: From Day 1 postoperative until discharge from PACU (up to 1 day)
Population: The outcome measure "total time in PACU" was not able to be assessed because there was no consistent measurement taken during the study by PACU nurses of this time period.
Arm/Group | Topical Lidocaine and Bupivacaine Alone | Topical Lidocaine and Bupivacaine With Thrombin | Topical Lidocaine and Bupivacaine With Thrombin and Tranexamic Acid | Topical Lidocaine and Bupivacaine With Thrombin and Aminocaproic Acid
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Topical Lidocaine and Bupivacaine Alone | Topical Lidocaine and Bupivacaine With Thrombin | Topical Lidocaine and Bupivacaine With Thrombin and Tranexamic Acid | Topical Lidocaine and Bupivacaine With Thrombin and Aminocaproic Acid
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT04814433/Prot_SAP_000.pdf